CLINICAL TRIAL: NCT04212533
Title: Vitamin D and Calcium Supplementation to Prevent Post-total Thyroidectomy Hypocalcaemia, a Comparative Clinical Trial
Brief Title: Preoperative Hypocalcaemia, a Comparative Clinical Trial
Acronym: professor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: hazem nour ca++
Record Dates: First submitted 2019-12-22; First posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Total Thyroidectomy
Keywords: hypocalcaemia, thyroidectomy, vit D, calcium
MeSH Terms: conditions — Hypocalcemia | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: two parallel groups each one 43 patients undergoing total thyroidectomy one received prophylactic vitamin d and calcium before surgery the other received nothing , calcium level, vit d levels measured preand postoperative , clinical assessment of patients postoperatie for development of tetany
Who Masked: Participant
Masking Description: the patients dont know what they received before the operation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supplementation arm (Active Comparator): 43 patients undergoing total thyroidectomy received 40000 IU vit D and once before operation and 500mg calcium tab 4 times in the day before surgery
  Interventions: Dietary Supplement: Vitamin D
- non-supplementation arm (Active Comparator): 43 patients undergoing total thyroidectomy received rice starch tablets /6 hrs in the day before surgery
  Interventions: Dietary Supplement: rice starch tablets

INTERVENTIONS:
Dietary Supplement: Vitamin D — comparison between pre- and postoperative calcium and vitamin d level after vit d and calcium supplementation
  Other Names: calcium supplementation
  Arms: supplementation arm
Dietary Supplement: rice starch tablets — rice starch tablets as placebo
  Arms: non-supplementation arm

SUMMARY:
two groups of patients undergoing total thyroidectomy one group received calcium and vit d prophylaxis the other group received no prophylaxis the investigator measured calcium level post and preoperative and development of tetant was recorded

DETAILED DESCRIPTION:
This study is randomized controlled trial carried out on 86 patients undergoing total thyroidectomy in the period between January 2018 and November 2019. Patients were randomly allocated into two groups each one 43 patients the first group is the supplementation group where patients received oral vitamin D 40000 IU and calcium tablets 1 g once before surgery.

Patient included in this study are those above 18 years old undergoing total thyroidectomy.

Patients excluded from this study are those with

* Previous thyroid surgery
* Malabsorption diseases
* Pregnancy
* Previous parathyroid disease or surgery
* Vitamin D deficiency
* Renal impairment
* Hypo or hyper calcaemia
* ASA class 3,4

all patients in this study were subjected to thorough history taking full clinical examination, body mass index calculation, proper assessment of the original thyroid disease requiring surgery, preoperative investigations done as usual in addition to serum calcium, serum magnesium, serum vitamin D and serum parathormon level.

Serum calcium and serum parathormon were tested after 6, 12 and 48 postoperative hours, patients were discharged on the third postoperative day except if further hospitalization was indicated, after discharge patients were followed up in the outpatient clinic by one of the surgical team, serum calcium and parathormon level were tested after1 months, 3 months and after 6th months.

The primary outcome of this study is the development of hypocalcaemia either clinically or laboratory.

Clinical hypocalcaemia means development of perioral and \ or acral tingling and numbness, twitches of the perioral region on tapping in front of the ear" Chvostec's sign'', muscle twitches and development of carpopedal spasm.

Laboratory hypocalcaemia means serum calcium level below 8.5 mg\dl. Secondary outcome is the postoperative parathormon level. Preoperative data, postoperative clinical follow up and laboratory data were collected and analyzed using SPSS 22 program package.

Principles of total thyroidectomy; Total thyroidectomy was performed under general anesthesia, through lower neck collar incision, skin and platysma muscle flap was raised till the thyroid cartilage, opening the midline raphe, exploration of each thyroid lobe and tracing the inferior thyroid artery while emerging from underneath the carotid artery, the inferior thyroid artery was identified with its branches supplying the parathyroid gland, which was identified and preserved with its blood supply, the recurrent laryngeal nerve was searched for in the triangle between the carotid artery , trachea and the inferior thyroid artery. The external laryngeal nerve was identified and preserved 1 cm superior to the upper thyroid pole. If radical thyroidectomy was deemed the same principles of preserving parathyroid glands and their blood supply, recurrent and external laryngeal nerves. If the surgeons ere sure of damaging or removing the parathyroid glands a half of one of them was minced and transplanted in the subcutaneous tissue of the left forearm

ELIGIBILITY:
Inclusion Criteria:

• patient undergoing total thyroidectomy

Exclusion Criteria:

* Previous thyroid surgery
* Malabsorption diseases
* Pregnancy
* Previous parathyroid disease or surgery
* Vitamin D deficiency
* Renal impairment
* Hypo or hyper calcaemia
* ASA class 3,4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
number of participants with hypocalcemia | 24 hrs post operative
  calcium level below 8.5 mg\dl measured by serum calcium assay
number of participants with hypocalcaemia | after 7 days post operative
  calcium level below 8.5 mg\dl measured by serum calcium assay

SECONDARY OUTCOMES:
number of participants with decreased parathormone level below normal level | ( 1st month post operative)
  level of parathormone below 10 pg/mL
number of participants with tetany | 1 week
  development of tingling, numbness or carpopedal spasm measured by clinical examination and patient history

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, Principal Investigator — zag university
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: No